CLINICAL TRIAL: NCT06897449
Title: The Effects of Positive Psychological Interventions on Identity,Mental Energy, Well-being, and Self- Compassion Among Chinese Collegiate Student-athletes
Brief Title: The Effects of Positive Psychological Interventions on Chinese Collegiate Student-athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Xiawei (Other)
Responsible Party: Sponsor-Investigator, Wang Xiawei, PHD student, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: USM/JEPeM/KK/23030250
Record Dates: First submitted 2024-11-01; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2023-07

CONDITIONS: Psychological Well-Being; Intervention
Keywords: student-athlete,unviersity
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Positive psychological intervention (Experimental): This experimental intervention is an eight-week positive psychology program aimed at enhancing student-athletes' identity, mental energy, well-being, and，self-compassion. The program guides participants through exercises such as recalling personal achievements, identifying character and athletic strengths, setting goals, and envisioning future aspirations. By fostering positive emotions, resilience, and connection with others, this intervention seeks to support athletes in achieving mental and emotional well-being, both in sports and in life.
  Interventions: Behavioral: Positive psychological intervention
- Introduction to Positive Psychology (Placebo Comparator): The control group intervention consists of an informational poster introducing positive psychology. This simple, non-interactive approach provides basic knowledge about positive psychology concepts without engaging participants in specific exercises or activities, serving as a minimal-intervention comparison for the active training program in the experimental group.
  Interventions: Other: Introduction to Positive Psychology Poster

INTERVENTIONS:
Behavioral: Positive psychological intervention — Each week consists of two modules, focusing on different techniques and methods from positive psychology, aimed at improving athletes' mental health and performance.
  Arms: Positive psychological intervention
Other: Introduction to Positive Psychology Poster — The poster serves as an introductory resource, summarizing key concepts of positive psychology in an accessible format.
  Arms: Introduction to Positive Psychology

SUMMARY:
The purpose of this study is to examine the effects of positive psychology intervention on the identity, psychological competence, well-being, and self-compassion of Chinese student-athletes. The first part of the study is guided by the theory of positive psychology and positive psychological interventions. Five scales, namely the Academic and Athletic Identity Scale, Athletic Mental Energy Scale, Sport Mental health Continuum-Short Form, Perceived Available Support in Sport Questionnaire, and Self-Compassion Scale-Short Form, are selected and translated from English into Chinese to validate the reliability and validity of the five scales in the Chinese population. The investigators will invite student-athlete to participate in a two-part study .This study will last approximately 8 weeks for a total of 12 interventions that have been shown to have a positive impact on people;s lives and the investigators would like to further examine the potential. participants will not be forced to participate in this study if they do not wish to.

DETAILED DESCRIPTION:
The experimental intervention is designed to enhance student-athletes' mental energy, well-being, self-compassion, and identity through an eight-week positive psychology training program. Each week consists of two modules, focusing on different techniques and methods from positive psychology, aimed at improving athletes' mental health and performance.

In Week 1, the intervention covers two modules: "Recreating Glory" and "Three Good Things." Participants will reflect on their personal achievements, write them down, and share these positive memories to enhance emotional regulation and self-awareness. The "Three Good Things" exercise encourages participants to recall three positive events each day, fostering positive thinking and broadening their perspective on life.

Week 2 focuses on "Sport Strengths" and "Character Strengths." Participants will identify their athletic strengths and areas for improvement, setting realistic goals to boost self-efficacy. They will also evaluate their character strengths with the help of family and friends, choosing the five that best represent them and reflecting on how these strengths shape their personal identity.

In Week 3, the modules "Using Strengths to Overcome Stress" and "Personal Growth Plan" will teach participants how to leverage their strengths to cope with stress and negative emotions. They will also develop a personal growth plan to envision a better future self, enhancing their well-being and goal achievement.

Week 4 includes "Positive Self-Talk" and "Optimistic Attribution." Participants will learn how to reduce self-criticism and increase self-esteem through compassionate self-talk. They will also be guided to attribute success and failure in a positive, rational way, helping them build resilience and confidence in handling unexpected challenges in sports.

In Week 5, the "Enjoying Life" module teaches participants how to slow down, focus on life's beauty, and relax. Music and mindful relaxation exercises are introduced to help them manage stress. Week 6, the "Acts of Kindness" module, encourages participants to use their strengths to help others, fostering a sense of accomplishment and emotional fulfillment through positive actions.

Week 7 focuses on "Positive Relationships," helping participants develop empathy and teamwork by recognizing the strengths of those around them, which enhances group cohesion. Lastly, in Week 8, the "Dream List" module prompts participants to think about and plan for their future aspirations, helping them pursue long-term goals and find meaning in life.

Overall, this intervention integrates various dimensions of positive psychology to promote comprehensive improvements in the mental energy, well-being, and self-awareness of student-athletes.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate student-athletes, who regularly train with their varsity sports teams
* Can represent the university at the University level and above
* 18 years old and above， informed and voluntary participation

Exclusion Criteria:

* Have a history of mental disorders and psychiatric illnesses
* Experienced a significantly stressful event, such as bereavement, loss of a loved one
* At risk of self-injury or suicide
* Participants who do not give their signed informed consent form will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in mental energy before and after the 8-Week positive psychological intervention | Baseline and 8 weeks after intervention.
  Mental energy levels will be assessed using the Athetic Mental Energy Scale (AMES), a validated tool for evaluating an individual's subjective perception of cognitive vigor, motivation, and alertness.The AMES consists of 18 items rated on a 6-point Likert scale. Higher scores reflect greater mental energy, while lower scores indicate mental fatigue or depletion.
Changes in identity after the 8-Week positive psychological intervention | Baseline and 8 weeks after intervention.
  Identity will be assessed before and after the 8-week positive psychological intervention. The measurement will be conducted using the Athletic and Acadmic identity Scale (AAIS). The AAIS evaluates the strength and exclusivity of an individual's identification with the athlete role.
Changes in Self-compassion Before and After the 8-Week Positive Psychological Intervention | Baseline and 8 weeks after intervention.
  Self-compassion will be measured using the Self-Compassion Scale (SCS), which assesses individuals' self-kindness, common humanity, and mindfulness in response to personal difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Xiawei Wang, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Positive Psychological Intervention, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No